CLINICAL TRIAL: NCT05777135
Title: Effect of Ringer Lactate Preloading on Induction Dose Requirement of Propofol and Its Haemodynamic Stability at a Tertiary Center
Brief Title: Ringer Lactate Preloading on Induction Dose Requirement of Propofol
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Medical College Birgunj (Other)
Responsible Party: Principal Investigator, Arushi Jaiswal, Postgraduate Doctor, National Medical College Birgunj
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 519 - 2022
Record Dates: First submitted 2023-02-01; First posted 2023-03-21 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-04

CONDITIONS: Anesthesia; Ringer's Lactate
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Preloading with Ringer Lactate) (Experimental): Preloading with Ringer lactate 30ml/kg over 30 minutes prior to surgery and Propofol dose requirement for induction of anaesthesia will be noted
  Interventions: Drug: Ringer Lactate prior to surgery and Propofol
- Group II (No preloading) (No Intervention): No preloading will be done and Propofol dose requirement for induction of anaesthesia will be noted

INTERVENTIONS:
Drug: Ringer Lactate prior to surgery and Propofol — Ringer Lactate prior to surgery and Propofol dose requirement for induction of anaesthesia will be noted
  Other Names: Ringer Lactate group
  Arms: Group I (Preloading with Ringer Lactate)

SUMMARY:
* To compare the effect (heart rate and mean arterial pressure) of Ringer Lactate preloading and without preloading on induction dose requirement of Propofol.
* The Propofol requirement for induction dose with respect to loss of eyelash reflex in Ringer Lactate preloaded versus control group.

DETAILED DESCRIPTION:
1. From the operation list, patients that meet the Inclusion criteria will be selected. (n=60)
2. Patients will be allocated into two participant groups. Group I and Group II respectively using Simple random sampling technique by Ballot method. Ballot method is to keep the list of patients that meet the inclusion criteria in two ballot box mentioning name and groups and do the lottery based selection for both groups and Patient code will be given.
3. Group I (n = 30) Preloading with Ringer Lactate 30 ml/kg over 30 mins prior to surgery will be done and Propofol dose (2mg / kg ) requirement for induction of anaesthesia will be noted.

   Group II (n = 30) No Preloading will be done and Propofol dose (2mg / kg) requirement for induction of anaesthesia will be noted.
4. Then, investigators will visualize for loss of eyelash reflex in both groups.
5. The hemodynamic response (heart rate, systolic blood pressure, diastolic blood pressure and mean arterial pressure) to intubation between the two participant groups will be noted. The total Propofol requirement for induction in Ringer Lactate preloaded versus control group will be recorded.
6. Drug administration and parameters recording will be done by the anaesthesiologist / under supervision

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for elective surgeries
2. American Society of Anaesthesiologists (ASA) class I patients
3. Age between 18-45 years
4. Any surgery under general anaesthesia requiring endotracheal intubation
5. Body mass index (BMI) -18.5 - 24.9
6. Those providing written consent

Exclusion Criteria:

1. Emergency surgery
2. Patients with multiple injuries, pregnancy
3. Airway Mallampati grade II, III and IV
4. Allergy to Ringer Lactate and Propofol.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Propofol dose Required (mg) | Standard dosing in Operation
  Propofol dose (mg) with aspect to weight (kg)
Total Propofol dose given (mg) | Visualization of loss of eyelash reflex
  Propofol dose (mg)
Loss of eyelash reflex (seconds) | Propofol given till loss of eyelash reflex
  Visualization of loss of eyelash reflex (seconds)

SECONDARY OUTCOMES:
Units of Measure (e.g., weight and height) | Preanaesthetic checkup, Day 1
  Weight in kilograms, height in meters ( weight and height will be combined to report BMI in kg/m²).
Heart rate (beats / minute): After IV Propofol | Immediately After IV Propofol
  Heart rate (beats / minute) will be measured with pulse oxymeter
Heart rate (beats / minute): Baseline before IV fluid infusion | Base line Before IV fluid infusion
  Heart rate (beats / minute) will be measured with pulse oxymeter
Heart rate (beats / minute): At intubation (0 minute) | At intubation (0 minute)
  Heart rate (beats / minute) will be measured with pulse oxymeter
Heart rate (beats / minute): Post intubation (1 minute) | Post intubation (1 minute)
  Heart rate (beats / minute) will be measured with pulse oxymeter
Heart rate (beats / minute): Post intubation (3 minute) | Post intubation (3 minute)
  Heart rate (beats / minute) will be measured with pulse oxymeter
Heart rate (beats / minute): Post intubation (5 minute) | Post intubation (5 minute)
  Heart rate (beats / minute) will be measured with pulse oxymeter
Heart rate (beats / minute): Post intubation (10 minute) | Post intubation (10 minute)
  Heart rate (beats / minute) will be measured with pulse oxymeter
Systolic blood pressure (mm Hg): Baseline before IV fluid infusion | Baseline before IV fluid infusion
  Systolic blood pressure (mm Hg) will be recorded on vital monitor
Systolic blood pressure (mm Hg): After IV Propofol | Immediately After IV Propofol
  Systolic blood pressure (mm Hg) will be recorded on vital monitor
Systolic blood pressure (mm Hg): At intubation (0 minute) | At intubation (0 minute)
  Systolic blood pressure (mm Hg) will be recorded on vital monitor
Systolic blood pressure (mm Hg): Post intubation (1 minute) | Post intubation (1 minute)
  Systolic blood pressure (mm Hg) will be recorded on vital monitor
Systolic blood pressure (mm Hg): Post intubation (3 minute) | Post intubation (3 minute)
  Systolic blood pressure (mm Hg) will be recorded on vital monitor
Systolic blood pressure (mm Hg): Post intubation (5 minute) | Post intubation (5 minute)
  Systolic blood pressure (mm Hg) will be recorded on vital monitor
Systolic blood pressure (mm Hg): Post intubation (10 minute) | Post intubation (10 minute)
  Systolic blood pressure (mm Hg) will be recorded on vital monitor
Diastolic blood pressure (mm Hg): Baseline before IV fluid infusion | Baseline before IV fluid infusion
  Diastolic blood pressure (mm Hg) will be recorded on vital monitor
Diastolic blood pressure (mm Hg): After IV Propofol | Immediately After IV Propofol
  Diastolic blood pressure (mm Hg) will be recorded on vital monitor
Diastolic blood pressure (mm Hg): At intubation (0 minute) | At intubation (0 minute)
  Diastolic blood pressure (mm Hg) will be recorded on vital monitor
Diastolic blood pressure (mm Hg): Post intubation (1 minute) | Post intubation (1 minute)
  Diastolic blood pressure (mm Hg) will be recorded on vital monitor
Diastolic blood pressure (mm Hg): Post intubation (3 minute) | Post intubation (3 minute)
  Diastolic blood pressure (mm Hg) will be recorded on vital monitor
Diastolic blood pressure (mm Hg): Post intubation (5 minute) | Post intubation (5 minute)
  Diastolic blood pressure (mm Hg) will be recorded on vital monitor
Diastolic blood pressure (mm Hg): Post intubation (10 minute) | Post intubation (10 minute)
  Diastolic blood pressure (mm Hg) will be recorded on vital monitor
Mean arterial pressure (mm Hg): After IV Propofol | Immediately After IV Propofol
  Diastolic blood pressure (mm Hg) will be recorded on vital monitor
Mean arterial pressure (mm Hg): Baseline before IV fluid infusion | Baseline before IV fluid infusion
  Diastolic blood pressure (mm Hg) will be recorded on vital monitor
Mean arterial pressure (mm Hg): At intubation (0 minute) | At intubation (0 minute)
  Diastolic blood pressure (mm Hg) will be recorded on vital monitor
Mean arterial pressure (mm Hg): Post intubation (1 minute) | Post intubation (1 minute)
  Diastolic blood pressure (mm Hg) will be recorded on vital monitor
Mean arterial pressure (mm Hg): Post intubation (3 minute) | Post intubation (3 minute)
  Diastolic blood pressure (mm Hg) will be recorded on vital monitor
Mean arterial pressure (mm Hg): Post intubation (5 minute) | Post intubation (5 minute)
  Diastolic blood pressure (mm Hg) will be recorded on vital monitor
Mean arterial pressure (mm Hg): Post intubation (10 minute) | Post intubation (10 minute)
  Diastolic blood pressure (mm Hg) will be recorded on vital monitor

CONTACTS AND LOCATIONS:
Locations (1):
- National Medical College Teaching Hospital, Birgunj, Madhesh, Nepal

REFERENCES:
- [Result] Smith I, White PF, Nathanson M, Gouldson R. Propofol. An update on its clinical use. Anesthesiology. 1994 Oct;81(4):1005-43. No abstract available. PMID 7943815
- [Result] Hug CC Jr, McLeskey CH, Nahrwold ML, Roizen MF, Stanley TH, Thisted RA, Walawander CA, White PF, Apfelbaum JL, Grasela TH, et al. Hemodynamic effects of propofol: data from over 25,000 patients. Anesth Analg. 1993 Oct;77(4 Suppl):S21-9. PMID 8214693
- [Result] Van Aken H, Meinshausen E, Prien T, Brussel T, Heinecke A, Lawin P. The influence of fentanyl and tracheal intubation on the hemodynamic effects of anesthesia induction with propofol/N2O in humans. Anesthesiology. 1988 Jan;68(1):157-63. doi: 10.1097/00000542-198801000-00031. No abstract available. PMID 3257362
- [Result] Briggs LP, Dundee JW, Bahar M, Clarke RS. Comparison of the effect of diisopropyl phenol (ICI 35, 868) and thiopentone on response to somatic pain. Br J Anaesth. 1982 Mar;54(3):307-11. doi: 10.1093/bja/54.3.307. PMID 6978144
- [Result] McCollum JS, Milligan KR, Dundee JW. The antiemetic action of propofol. Anaesthesia. 1988 Mar;43(3):239-40. doi: 10.1111/j.1365-2044.1988.tb05551.x. PMID 3259081
- [Result] Williams EL, Hildebrand KL, McCormick SA, Bedel MJ. The effect of intravenous lactated Ringer's solution versus 0.9% sodium chloride solution on serum osmolality in human volunteers. Anesth Analg. 1999 May;88(5):999-1003. doi: 10.1097/00000539-199905000-00006. PMID 10320158